CLINICAL TRIAL: NCT05558761
Title: Clinical Study to Evaluate the Possible Efficacy of Pentoxifylline in Patients With Ulcerative Colitis Treated With Mesalamine
Brief Title: Pentoxifylline as Adjunctive Therapy in Patients With Ulcerative Colitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mostafa Bahaa, Teaching Assistant, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3455
Record Dates: First submitted 2022-09-25; First posted 2022-09-28 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases | interventions — Pentoxifylline

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: double-blinded
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): this group will take mesalamine 1 g three times daily
- Pentoxifylline group (Active Comparator): his group will take mesalamine 1 g three times daily plus pentoxifylline 400 mg two times daily
  Interventions: Drug: Pentoxifylline 400 MG

INTERVENTIONS:
Drug: Pentoxifylline 400 MG — Pentoxifylline (PTX) is a methyl-xanthine derivative that possesses antioxidant and anti-inflammatory characteristics. PTX exerts anti-inflammatory effects by inhibiting phosphodiesterase and activating the adenosine 2 receptor
  Arms: Pentoxifylline group

SUMMARY:
The exact underlying mechanisms of ulcerative colitis (UC), an idiopathic, chronic inflammatory disease marked by diffused inflammation of the colon and rectum mucosa, are still unknown. Due to genetic, immune, and environmental factors, UC is highly dependent on cellular immune reactions and exaggerated inflammatory responses. The release of several cytokines, kinins, leukotrienes, platelet-activating factor (PAF), and reactive oxygen species is connected to immunological activity (ROS). Additionally, many of the cytokines will start an acute phase response, making the inflammation worse.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years Both males and females will be included Negative pregnancy test and effective contraception

Exclusion Criteria:

- Breastfeeding Significant liver and kidney function abnormalities Colorectal cancer patients Patients with severe UC Patients taking rectal or systemic steroids Known allergy to the studied medications

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-10-10 (Actual); Primary Completion 2024-04-20 (Actual); Study Completion 2024-04-20 (Actual)

PRIMARY OUTCOMES:
Improvement in health related quality of life | 6 months
  Short Form 36 Health Survey (SF-36) will assess the quality of life. The SF-36 is an indicator of overall health status and contains 10 items. The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100. Lower scores = more disability, higher scores = less disability

SECONDARY OUTCOMES:
changes in the level of measured biomarkers. | 6 months
  changes in the level of measured biomarkers through assessment serum level of TNF- alpha, serum IL-10, and gene expression of zonula occuldin-1(ZO-1).

CONTACTS AND LOCATIONS:
Overall Officials: Mostafa M Bahaa, PhD, Principal Investigator — Pharmacy Practice Department, Faculty of Pharmacy, Horus University, New Damietta, Egypt
Locations (1):
- Faculty of Medicine, Mansoura University, Al Mansurah, Egypt

REFERENCES:
- [Derived] Bahaa MM, Hegazy SK, Maher MM, Bahgat MM, El-Haggar SM. Pentoxifylline in patients with ulcerative colitis treated with mesalamine by modulation of IL-6/STAT3, ZO-1, and S1P pathways: a randomized controlled double-blinded study. Inflammopharmacology. 2024 Oct;32(5):3247-3258. doi: 10.1007/s10787-024-01560-6. Epub 2024 Aug 27. PMID 39192162